CLINICAL TRIAL: NCT05958082
Title: Utilization of Educational Interventions in Completion of Genetic Testing in Black Patients With High-Risk Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Clara Hwang, Principal Investigator, Clinical Assistant Professor, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 16491; HFH-23-01 (Other: Henry Ford CCTRO)
Record Dates: First submitted 2023-07-07; First posted 2023-07-24 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: genetic testing
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational intervention (Experimental): Patients will be asked questions about genetic testing for prostate cancer before and after an educational intervention.
  Interventions: Behavioral: Educational video

INTERVENTIONS:
Behavioral: Educational video — The educational intervention will occur with a clinical research coordinator who will be trained to educate on germline testing in prostate cancer.

SUMMARY:
This is a pilot study to improve rates of germline genetic testing for black patients with aggressive prostate cancer as recommended by the updated guidelines by the National Cancer Comprehensive Network (NCCN) in 2018.

In this study, consented patients will undergo a low-risk intervention of an educational session with a trained staff member on germline testing in prostate cancer and, if agreeable, subsequent germline cancer genetic testing via a commercial lab test.

DETAILED DESCRIPTION:
This is a prospective, single-arm, quality improvement initiative for the use of a standardized educational intervention on germline testing in black patients with prostate cancer to improve the rates of germline genetic testing among those recommended for testing. Patients who consent to the study will undergo a one-on-one in-person education session regarding the rationale and the benefits/risks of germline testing.

The educational intervention will occur with a clinical research coordinator who will be trained to educate on germline testing in prostate cancer. At the start of the session, the patient will be given a short questionnaire to assess their understanding about germline and genetic testing, along with a Family History questionnaire.

Following the educational intervention, the patient will be asked to complete a short patient education and satisfaction questionnaire.

If a patient wishes to proceed with testing, they will sign the standard consent to proceed with germline testing via a commercial assay. Upon a patient deciding to pursue testing, testing will consist of a prostate cancer germline panel with a commercially available blood or saliva-based assay. Upon receipt of the results, the coordinator will alert the patient's clinician, who will then share the results with the patient either in clinic or by phone. If the results show a pathogenic germline mutation, the patient will be referred to see Henry Ford Health genetics clinic for consultation with a genetics counselor.

If a patient pursues genetic testing, following receipt of results, the patient's clinicians will be asked to complete a short survey on to assess how the results of germline testing affected the patient's current and future management.

ELIGIBILITY:
Inclusion Criteria:

1. Men, age greater than or equal to 18 years of age.
2. Men who racially identify as black or multiracial including black
3. Diagnosis of prostate cancer of any histology.
4. Must meet NCCN guidelines for germline testing

   1. Men with very low, low or intermediate risk prostate per NCCN guidelines with a positive family history or intraductal histology. Family history here is considered significant if the patient has:

      * a first degree relative with prostate cancer or more than one first/second degree relative with prostate cancer, or
      * ≥3 cancers on same side of family, especially diagnoses ≤50 years of age: bile duct, breast, colorectal, endometrial, gastric, kidney, melanoma, ovarian, pancreatic, prostate (but not clinically localized Grade Group 1), small bowel, or urothelial cancer
   2. Men with high-risk, very-high risk (per NCCN definitions of risk groups), lymph node positive, or metastatic prostate cancer independent of family history of histology.

Exclusion Criteria:

1. Have had prior germline testing.
2. Have somatic genetic testing that is positive for a possible germline variant.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Testing rate | 24 months
  percentage of patients who undergo genetic testing after completing the education session

SECONDARY OUTCOMES:
Baseline knowledge per "Patient Survey on Germline Testing in Prostate Cancer" questionnaire | Day 1, before intervention
  Pre-Intervention Patient Questionnaire: The pre-intervention patient questionnaire is a brief 16-item investigator-developed knowledge and attitude scale applicable to this population. It was developed through an expert panel to determine if participants are able to recall key core components about multigene panel testing and capture attitudes about genetic testing. This survey is estimated to take 10 minutes to complete.
Post-intervention knowledge per "Patient Post-Education Patient Survey" questionnaire | Day 1, after intervention
  Post-Intervention Patient Questionnaire: The post-intervention patient questionnaire is a brief 24-item investigator-developed knowledge and attitude scale applicable to this population. It includes the same 14 knowledge and attitude items from the pre-intervention survey to assess impact of the educational intervention. It was developed through an expert panel to determine if participants are able to recall key core components about multi-gene panel testing and capture attitudes about genetic testing. There is also a 10-item scale to capture satisfaction with educational intervention. This survey is estimated to take 10 minutes to complete.
Clinician attitudes per "Post Results Clinician Questionnaire" | 24 months
  Post-Results Clinician Questionnaire: The post-result clinician questionnaire is a brief 6-item investigator-developed scale to assess whether the genetic testing results altered clinical practice for any given patient including change in disease monitoring, change in recommended treatment, referral to genetic counseling and other parameters. This survey is estimated to take 5 minutes to complete.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Cancer Pavilion, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No